CLINICAL TRIAL: NCT00451672
Title: The Therapeutic Effect of Bromocriptin in Patients With Primary Aldosteronism
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 950912
Expanded Access: Available
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2007-03-23 (Estimated); Status verified 2006-12

CONDITIONS: Hyperaldosteronism; Hypertension
Keywords: aldosteronism, bromocriptin, hypertension
MeSH Terms: conditions — Hyperaldosteronism; Hypertension | interventions — Bromocriptine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: bromocriptine

SUMMARY:
we propose that bromocriptine may be an alternative treatment of primary aldosteronism, both APA and BAH.

DETAILED DESCRIPTION:
Primary aldosteronism (PA), a common curable disease of hypertension, is characterized by inappropriate production of aldosterone, which is at least partially autonomous of the renin-angiotensin system. A recent clinical study reported that patients with PA experience a higher sate of a higher rate of cardiovascular events than those with essential hypertension(Corry and Tuck 2003; Milliez, Girerd et al. 2005). The prevalence of metabolic syndrome was higher in primary aldosteronism than in essential hypertension was also reported (Fallo, Veglio et al. 2006). The wide applying of the plasma aldosterone/plasma rennin activity (ARR) as a screening test among hypertensive patients have reported a much higher prevalence of this disease, up to 12% of hypertensive patients. In the past decade, an increase in diagnosis rate of PA has been observed in National Taiwan University Hospital, with an average of 15-20 newly diagnosis cases every year.

Idiopathic bilateral adrenal hyperplasia (BAH) and aldosterone-producing adenoma (APA) are the leading causes of primary aldosteronism. Unilateral adrenalectomy is the reasonable therapeutic option of APA and aldosterone antagonists usually brings about well blood pressure (BP) control in BAH. Not every APA patient would accept operation because of other medical conditions, or the cure rate of hypertension in APA after adrenalectomy is 50-70% in most studies. For patients with BAH, aldosterone antagonists are the first choice of treatment, however, intolerance to high dose of these medications is not uncommon. To our best knowledge, there is no alternative treatment for these patients.

Dopaminergic regulation of aldosterone secretion has been well demonstrated in normal subjects as well as patients with PA. We have shown that D2 receptor can down-regulate the transcription of aldosterone synthase (CYP11B2) via a specific PKC isoform and probably intracellular calcium level. Furthermore, there is a reciprocal change of the mRNA of D2 receptor and CYP11B2 in APA. D2 receptor has also been demonstrated in other neuroendocrine tumors, eg., pheochromocytoma, prolactinoma, GH-secreting adenoma ect. [Camacho & Mazzone 1999] Administration of D2 agonist, bromocriptin (BMC), is a standard treatment of prolactinoma, either for pre-operative reduction of the tumors or for non-surgical patients [Chattopadhyay et al., 2005]. Reduction or shrinkage of prolactinoma has been observed in patients treated with BMC [Biswas et al., 2005]. Anti-proliferative effect and apoptosis of BMC have been demonstrated in several cell lines [Wasko et al., 2004]. Recently, we also demonstrated that BMC, in addition to decrease aldosterone secretion and expression of CYP11B2, could inhibit cell proliferation of H295 cells, an adrenocortical carcinoma cell line, with a down-regulation of ERK. In this context, we propose that BMC may be an alternative treatment of PA, both APA and BAH.

ELIGIBILITY:
Inclusion Criteria:

* 20-60y/o hyperaldosteronsim patients

Exclusion Criteria:

* Malignancy
* Bed-ridden
* Psychological disease

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25
Dates: Start 2007-01; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
tumor size, blood pressure

SECONDARY OUTCOMES:
serum potassium, aldosterone, renine

CONTACTS AND LOCATIONS:
Overall Officials: Kwan-Dun Wu, MD, PhD, Principal Investigator — Internal Medicine, Natinal Taiwan University Hospital; Vin-Cent Wu, MD, Study Director — Internal Medicine, National Taiwan University Hospital
Locations (1):
- National Taiwan Univserty Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Chang HW, Chu TS, Huang HY, Chueh SC, Wu VC, Chen YM, Hsieh BS, Wu KD. Down-regulation of D2 dopamine receptor and increased protein kinase Cmu phosphorylation in aldosterone-producing adenoma play roles in aldosterone overproduction. J Clin Endocrinol Metab. 2007 May;92(5):1863-70. doi: 10.1210/jc.2006-2338. Epub 2007 Feb 13. PMID 17299068